CLINICAL TRIAL: NCT06749808
Title: A Randomized, Double-Blind, Placebo Controlled, Single Center Study to Assess the Impact of a Nutritional Supplement on Wellbeing and Nutrient Absorption
Brief Title: A Study to Assess the Impact of a Nutritional Supplement on Wellbeing and Nutrient Absorption
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NSE-66-24
Record Dates: First submitted 2024-12-13; First posted 2024-12-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Nutrition Status
Keywords: carotenoids; nutritional supplement; nutritional status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Carotenoid Nutritional Supplement: capsules with 500 mg Vitamin C, 200 IU Vitamin E, 25 mg Zinc, 2 mg Copper, 70 mcg Selenium, 10 mg Lutein, 2 mg Zeaxanthin, 3mg boron, 255mg calcium, 100mcg chromium, 0.9mg copper, 150mcg iodide, 180mg magnesium, 75mcg molybdenum, 2.3mg manganese, 140mcg selenium, 20mcg vanadium, 15mg zinc
  Interventions: Dietary Supplement: Carotenoid Nutritional Supplement
- Placebo (Placebo Comparator): Placebo Supplement: capsules with 500 mg Vitamin C, 200 IU Vitamin E, 25 mg Zinc, 2 mg Copper, 70 mcg Selenium, 3mg boron, 255mg calcium, 100mcg chromium, 0.9mg copper, 150mcg iodide, 180mg magnesium, 75mcg molybdenum, 2.3mg manganese, 140mcg selenium, 20mcg vanadium, 15mg zinc
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carotenoid Nutritional Supplement — Carotenoid Nutritional Supplement: capsules with 500 mg Vitamin C, 200 IU Vitamin E, 25 mg Zinc, 2 mg Copper, 70 mcg Selenium, 10 mg Lutein, 2 mg Zeaxanthin, 3mg boron, 255mg calcium, 100mcg chromium, 0.9mg copper, 150mcg iodide, 180mg magnesium, 75mcg molybdenum, 2.3mg manganese, 140mcg selenium, 20mcg vanadium, 15mg zinc
  Arms: Active
Dietary Supplement: Placebo — Placebo Supplement: capsules with 500 mg Vitamin C, 200 IU Vitamin E, 25 mg Zinc, 2 mg Copper, 70 mcg Selenium, 3mg boron, 255mg calcium, 100mcg chromium, 0.9mg copper, 150mcg iodide, 180mg magnesium, 75mcg molybdenum, 2.3mg manganese, 140mcg selenium, 20mcg vanadium, 15mg zinc
  Arms: Placebo

SUMMARY:
The objective of this placebo controlled randomized research is to demonstrate the health benefits of a carotenoid nutritional supplement as compared to placebo in terms of nutrient levels, quality of life, feelings, of wellness, brain health, energy, immunity, and appearance.

DETAILED DESCRIPTION:
Female or male subjects will be enrolled in this single site study to evaluate the efficacy and tolerability of a nutritional supplement. Subjects who sign consent and meet all inclusion criteria and none of the exclusion criteria will be enrolled at the baseline visit. Vital signs will be obtained (height, weight, blood pressure, heart rate). Subjects must meet the study BMI requirements (≥18.5 and ≤29.9 kg/m2 ). Subjects will also complete BioPhotonic Scanner screening. If subjects meet all requirements, they will be randomized to receive either the active nutritional supplement or a placebo. Subjects will undergo phlebotomy for baseline lab work consisting of carotenoid analysis. Subjects will complete the following questionnaires/measurements:

1. Quality of Life Questionnaire
2. Diet and Lifestyle Questionnaire
3. Subject Skin Assessment
4. Biophotonic Scanner measurement
5. Mini-4 Scanner measurement

The nutritional supplement will be started and the subjects will return to the research center at Weeks 4 and 8 for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects male or female age 20-65 years old.
2. Subjects who score 30,000 or below on the Pharmanex BioPhotonic Scanner.
3. Subjects of Fitzpatrick skin types I-VI with no known medical conditions that, in the investigator's opinion, may interfere with study participation.
4. Subjects must be able to read, understand and provide written informed consent.
5. Individuals must agree to continue to use all regular brands of cosmetics and the assigned test materials for the duration of the study. Individuals must refrain from using any new products other than the assigned test supplements.
6. Subjects must agree to avoid excessive sun exposure (no more than 10-15 minutes of direct sunlight without SPF protection) and the use of artificial tanning methods for the duration of the study.

   -

Exclusion Criteria:

* 1. Individuals who are participating in any other research study. 2. Subjects who are regularly taking oral nutritional supplements containing carotenoids as specified by the sponsor.

  3. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study supplement.

  4. Concurrent therapy with any medication either topical or oral that might interfere with the study.

  5. Subjects who are alcohol or narcotic addicts. 6. Subjects who are unwilling to leave their current oral medications unchanged for the duration of the study.

  7. Subjects who use an indoor tanning booth. 8. Subjects, who are pregnant, breast feeding or planning a pregnancy. 9. Subjects with clinically significant unstable medical disorders, such as cancer, diabetes, neurodegenerative disorders, active autoimmune disease, liver or kidney disease, schizophrenia, depression, other major mental illness.

  10. Subjects who are cigarette smokers. 11. Subjects who regularly use supplements containing >2mg carotenoids such as: LifePak, Beauty Focus Collagen+, ageLOC Youth.

  12. Subjects who are unwilling or unable to comply with the requirements of the protocol.

  13. Subjects who are participating in another similar research study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Nutrient analysis | 8 weeks
  Nutrient levels as measured by blood serum carotenoids and correlated to BioPhotonic Scanner and Mini-4 scanner assessment. Higher blood serum carotenoid levels and scan scores indicate greater improvement.
Wellness Assessment | 8 weeks
  Subject self-assessment of global wellness via questionnaire. Likert Scale: 1=Strongly Disagree, 2=Disagree, 3=Neutral, 4=Agree, 5=Strongly Agree. Higher score indicates greater satisfaction/improvement.

SECONDARY OUTCOMES:
Skin Attribute Assessment | 8 weeks
  Assessment of facial skin improvements evaluated by self-perception questionnaire. Likert Scale: 1=Strongly Disagree, 2=Disagree, 3=Neutral, 4=Agree, 5=Strongly Agree. Higher scores indicate greater satisfaction/improvement.
Product Safety | 8 weeks
  Adverse event monitoring. Self-reported to primary investigator and documented.
Product Safety | 8 weeks
  Weight (in kg) will be recorded to calculate for BMI (kg/m^2).
Product Safety | 8 weeks
  Height: will be recorded in meters to used in BMI calculations (kg/m^2).

CONTACTS AND LOCATIONS:
Locations (1):
- Nu Skin, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No